CLINICAL TRIAL: NCT04873752
Title: An Exploratory Study to Investigate the Safety and Efficacy of UC-MSCs in Pediatric Patients With Cerebral Palsy
Brief Title: A Study to Investigate the Safety and Efficacy of UC-MSCs in Pediatric Patients With Cerebral Palsy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rohto Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UDI-001-0555
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Palsy; Periventricular Leukomalacia
MeSH Terms: conditions — Cerebral Palsy; Leukomalacia, Periventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- UDI-001 (Experimental): Four cycles with 8 administrations
  Interventions: Biological: UDI-001

INTERVENTIONS:
Biological: UDI-001 — 2.5 x 10^6 cells/kg of UDI-001 are administered intravenously. One cycle consists of twice a week administrations.

SUMMARY:
UDI-001 is administered to pediatric patients with cerebral palsy attributed to periventricular leukomalacia (PVL) multiple times to investigate its safety and efficacy.

DETAILED DESCRIPTION:
This is the first study of UDI-001 to be administered to children. Pediatric patients with cerebral palsy attributed to PVL are enrolled to the study and umbilical cord derived mesenchymal stromal cells (UC-MSCs) are administered to those patients multiple times intravenously. Safety and efficacy of UC-MSCs are evaluated for 52 weeks after the first administration.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 12 months and < 24 months corrected age at the time of informed consent
* Diagnosed with cerebral palsy
* Diagnosed with PVL
* GMFCS level between II and IV
* Able to obtain written informed consent from parents (legal representative)

Exclusion Criteria:

* Presence of progressive neurological disease
* Presence of congenital anomaly
* Diagnosed with Grade 3 or more severe intraventricular hemorrhage
* Body weight < 5kg
* Profound intellectual disorder
* Complication of serious infection such as sepsis
* Requirement of mechanical ventilation
* Complication of serious organ failure such as kidney, liver or heart diseases or others and considered to be inappropriate
* Diagnosed with or suspected of hypsarrhythmia
* Positive for HBV, HCV, HIV or HTLV-1
* Patients who have received cell therapy
* Patients who have undergone selective dorsal rhizotomy or received botulinum toxin products within a certain period of time

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Safety: Adverse Event | until Week 52
  Adverse events which appear in the participants after the treatment

SECONDARY OUTCOMES:
Gross Motor Function Measure Score (GMFM Score) | baseline to Week 52
  Difference and change in GMFM score
Gross Motor Function Classification System (GMFCS) | baseline to Week 52
  Improvement rate of GMFCS
Function Independence Measure for Children (WeeFIM) | baseline to Week 52
  Change in WeeFIM score
Kyoto Scale of Psychological Development Test 2001 (KSPD) | baseline to Week 52
  Change in and Improvement rate of KSPD

CONTACTS AND LOCATIONS:
Overall Officials: Sumito Okawa, Study Director — Rohto Pharmaceutical Co., Ltd.
Locations (1):
- Osaka City University Hospital, Osaka, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No